CLINICAL TRIAL: NCT01403337
Title: Cardiac Remote Ischemic Preconditioning Before Elective Major Vascular Surgery (CRIPES)
Brief Title: Cardiac Remote Ischemic Preconditioning Before Elective Major Vascular Surgery
Acronym: CRIPES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Veterans Research and Education (Other)
Responsible Party: Principal Investigator, Santiago Garcia, Staff Cardiologist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 411652941
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; myocardial infarction
MeSH Terms: conditions — Peripheral Arterial Disease; Myocardial Infarction | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Blood pressure cuff inflated in the right or left arm to 40-50 mmHg
  Interventions: Other: Control
- Preconditioning (Active Comparator): The RIPC protocol will consist of three cycles of the following: 5-minute inflation of a blood pressure cuff around the right upper arm to 200 mmHg (or 20 above the systolic blood pressure if baseline BP > 200 mmHg) to allow for external compression of the brachial artery resulting in transient arm ischemia, followed by a 5-minute interval of cuff deflation to allow for reperfusion. The total duration of the protocol is 30 minutes equally divided between ischemia and reperfusion. The protocol is to be applied in the patient room the morning of the operation.
  Interventions: Other: Ischemic preconditioning

INTERVENTIONS:
Other: Ischemic preconditioning — The RIPC protocol will consist of three cycles of the following: 5-minute inflation of a blood pressure cuff around the right upper arm to 200 mmHg (or 20 above the systolic blood pressure if baseline BP > 200 mmHg) to allow for external compression of the brachial artery resulting in transient arm ischemia, followed by a 5-minute interval of cuff deflation to allow for reperfusion. The total duration of the protocol is 30 minutes equally divided between ischemia and reperfusion. The protocol is to be applied in the patient room the morning of the operation.
  Arms: Preconditioning
Other: Control — A Blood Pressure cuff inflated to 40-50 mmHg
  Arms: Control

SUMMARY:
Vascular surgery is considered a high-risk operation with an anticipated risk of major cardiovascular complications in excess of 5%. The occurrence of a cardiovascular complication after surgery carries a long-term higher mortality risk. The main objective of this investigation is to reduce the proportion of patients having major cardiovascular complications during surgery through a clinical protocol of remote preconditioning that is safe, effective and reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients would be those undergoing elective major vascular surgery at the Minneapolis VA Medical Center for an expanding abdominal aortic aneurysm, obstructive carotid disease, and/or chronic limb ischemia during the study period. All patients must be ≥ 18 years of age and provide written informed consent.

Exclusion Criteria:

* Exclusion criteria include hypertensive crisis, acute coronary syndrome in the preceding 6 weeks, severe valvular heart disease, peripheral arterial disease of the upper extremities, manifested by a systolic blood pressure difference greater than 20 mmHg, pregnant women, patients unable to understand the consent process due to mental illness, advanced malignancy with limited life expectancy (<1 year), and hemodialysis with a fistula in the upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Troponin I elevation above the URL | Within 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Garcia, MD, Principal Investigator — Minneapolis VA Medical Center and The University of Minnesota
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States